CLINICAL TRIAL: NCT04402593
Title: Music Therapy For The Treatment Of Cisplatin Induced Tinnitus In Patients With Relapsed Germ Cell Cancer (rGCC): A Pilot Study
Brief Title: Music Therapy For The Treatment Of Cisplatin Induced Tinnitus In Patients With rGCC: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to staffing changes and no potential subjects at this time.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Debra S. Burns, Chair of the Department of Music and Arts Technology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCC-0673
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Relapsed Germ Cell Cancer; Cisplatin Induced Tinnitus
Keywords: relapsed germ cell cancer; cisplatin induced tinnitus; music therapy; germ cell cancer
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Intervention Model Description: Study will enroll 15 subjects to a twice a week Music Therapy intervention (modified Heidelberg Model of Neuro-Music Therapy) for 3 weeks (6 sessions total).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Heidelberg Model of Neuro-Music Therapy (mHNMT) (Experimental): The mHNMT for Tinnitus program was modified based on participant feedback of the original HNMT. This study will include 6 sessions, 2 sessions a week including the following interventions: resonance training, music relaxation, Intonation Training and session review/homework.
  Interventions: Behavioral: Modified Heidelberg Model of Neuro-Music Therapy

INTERVENTIONS:
Behavioral: Modified Heidelberg Model of Neuro-Music Therapy — 6 sessions, 2 sessions a week including the following interventions: resonance training, music relaxation, Intonation Training and session review/homework.

SUMMARY:
Pilot study evaluating the feasibility of recruitment, retention, and compliance to a modified Heidelberg Model of Neuro-Music Therapy (mHNMT) in patients with Cisplatin-induced Tinnitus and relapsed Germ Cell Cancer (rGCC).

DETAILED DESCRIPTION:
This is a prospective, interventional pilot study that plans to enroll 15 patients who are receiving salvage high dose chemo and bone marrow transplant for relapsed Germ cell Cancer (rGCC). Patients will be asked to go through a series of surveys and screening procedures to determine eligibility. Once enrolled, patients will receive music therapy while they are being treated either inpatient or outpatient for their standard of care treatments.

Primary Objective To evaluate the feasibility of recruitment, retention, and compliance to a mHNMT in patients with CIT and rGCC admitted to BMT service to undergo salvage high-dose chemotherapy with tandem bone marrow rescue.

Secondary Objectives To estimate the effects of mHNMT on severity of CIT, associated distress, anxiety, depression, fatigue, benefit findings, sleep, and audiometry measures and assess number of times homework completed.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent.
2. English speaking.
3. Ability to provide written informed consent and HIPAA authorization
4. Confirmed diagnosis of CIT via a score on the TFI of 26 or greater.
5. Personal history of rGCC.
6. Previous exposure to cisplatin.
7. Admitted to BMT service to undergo HDC-tBMR for the first time. (Because this is a feasibility study, a minimum number of MT sessions will not be required).
8. Agrees not to receive music therapy outside of study.

Exclusion Criteria:

1. Severe hearing impairment greater than 60 dB HL in the region of the center tinnitus frequency
2. Patient's tinnitus can not be pitch matched.
3. Clinical diagnosis of severe mental disorder or psychiatric or neurological disease such as psychosis, epilepsy, Parkinson's disease, dementia, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 30 days
  The ability to enroll at least 50% of approached subjects.
Retention feasibility | from the start of intervention until last subject completes intervention (i.e. up to 2 years)
  The ability to successfully retain 60% of enrolled subjects.
Compliance and fidelity feasibility | from the start of intervention until last subject completes intervention (i.e. up to 2 years)
  The ability to deliver over 90% of planned intervention.

SECONDARY OUTCOMES:
Effects of intervention on severity of Cisplatin Induced Tinnitus determined by scores on the Tinnitus Functional Index | Baseline, day +50, day +100, and day +270
  The Tinnitus Functional Index (TFI) has eight subscales that address the intrusiveness of tinnitus, the sense of control the patient has, cognitive interference, sleep disturbance, auditory issues, relaxation issues, quality of life, and emotional distress. Minimum value is 1 and maximum value is 10. A higher score indicates worse tinnitus.
  A mean score of 25 or less than 25 indicates relatively mild tinnitus and little or need for intervention. A mean score ranging from 25-50 indicates significant problems with tinnitus and a possible need for intervention. A mean score of 50 or greater indicates tinnitus severe enough to qualify for more aggressive intervention.
Effects of intervention on associated distress determined by scores on the Tinnitus Questionnaire | Baseline, day +50, day +100, and day +270
  For each item, individuals indicate the level of agreement by answering; not true (score 0), partly true (score 1), or true (score 2). A three point scale limits its utility as an outcome measure. Total scores range from 0-82, with higher scores indicating more distressing tinnitus.
Effects of intervention on anxiety determined by scores on the Impact of Events Scale | Baseline, day +50, day +100, and day +270
  A 22-item self-report measure that assesses subjective distress caused by traumatic events on a scale from 0-4, where 0 is not at all, and 4 is extremely. A higher score indicates increased anxiety.
Effects of intervention on depression determined by scores on Hospital Anxiety and Depression Scale | Baseline, day +50, day +100, and day +270
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal.
Effects of intervention on benefit findings determined by scores on The Benefit Finding Scale | Baseline, day +50, day +100, and day +270
  Uses a 5-point Likert scoring method from 1 = Not at all to 5 = Extremely.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Adult Short Form | Baseline, day +50, day +100, and day +270
  Use a 5-point Likert scale and employ 7-day recall. Higher scores indicate higher levels of fatigue. Scores are standardized (M = 50, SD = 10)
Number of hours asleep | Up to 3 weeks
  Actiwatch Spectrum Pro watch. Sleep parameters will be computed using Actiware® software. The sleep parameters produced include total sleep time, sleep latency (minutes until sleep onset), sleep efficiency, frequency and duration of awakenings after sleep onset (WASO), and number of awakenings. These Sleep variables will be scored for each 24-hour period, and averages over the course of use will be computed for nighttime sleep alone and nighttime sleep plus daytime naps to be combined into epochs for assessment.
Number of times homework completed | Each day of intervention until study completion, about 3 weeks
  This will be assessed each day of the intervention and captured using the Actiwatch Spectrum Pro and summed over the entire intervention period.
Audiometric evaluation | Baseline and day +270 (+/- 90 days)
  The Pure-tone hearing threshold audiometry (PTA) measures and classifies hearing loss into three levels: <25 dB (normal hearing); ≥25 dB <40 dB (mild hearing impairment); and ≥40 dB (moderate-to-severe hearing impairment). PTA will be measured in a soundproofing booth using an audiometer (SA 203, Entomed, Sweden), and include frequencies of 500, 1000, 2000, 3000, 4000, and 6000 Hz in both ears in accordance with the American National Standards Institute (ANSI) standard. The hearing threshold will be defined as the mean hearing threshold of the better ear on PTA tests at 500, 1000, 2000, and 4000 Hz. Hearing loss in this study will be defined as follows: <25 dB (normal hearing), ≥25 dB and <40 dB (mild hearing loss), and ≥40 dB (moderate-to-severe hearing loss).

CONTACTS AND LOCATIONS:
Overall Officials: Debra Burns, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States